CLINICAL TRIAL: NCT06671275
Title: A Single-arm, Open-label, Dose-escalation Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Preliminary Efficacy of CUD005 Injection in Patients with Liver Cirrhosis
Brief Title: A Clinical Study to Evaluate CUD005 Injection in Patients with Liver Cirrhosis
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KDS-CUD
Record Dates: First submitted 2024-08-25; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Cirrhosis Liver
Keywords: macrophage; Cirrhosis; cell therapy; PBMC; safety; tolerability; MTD; DLT; dose escalation
MeSH Terms: conditions — Fibrosis | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm cell therapy (Experimental): The study was designed according to the 3+3 principle, with a total of 3 dose levels and dose escalation.
  Low-dose group: 5.0×107 cells/time; Medium-dose group: 1.5×108 cells/time; High-dose group: 5.0×108 cells/time. Subjects were sequentially placed in 3 different dose groups administered as a single peripheral intravenous dose.
  According to the enrollment restriction design, a total of a minimum of 9 subjects are expected to be enrolled, and the final sample size depends on the number of DLT, the number of dose groups ascended before DLT is observed, and the MTD is determined.
  Interventions: Biological: Cell therapy

INTERVENTIONS:
Biological: Cell therapy — Subjects were placed sequentially into three different dose groups, 5.0×107 cells/time (low-dose group), 1.5×108 cells/time (medium-dose group), and 5.0×108 cells/time (high-dose group) for dose escalation

SUMMARY:
A single-arm, open-label, dose-escalation phase I clinical trial to evaluate the safety, tolerability, and preliminary efficacy of CUD005 injection in patients with liver cirrhosis

DETAILED DESCRIPTION:
The study was designed according to the 3+3 principle, with a total of 3 dose levels and dose escalation.

Low-dose group: 5.0×107 cells/time; Medium-dose group: 1.5×108 cells/time; High-dose group: 5.0×108 cells/time. Subjects were sequentially placed in 3 different dose groups administered as a single peripheral intravenous dose.

According to the enrollment restriction design, a total of a minimum of 9 subjects are expected to be enrolled, and the final sample size depends on the number of DLT, the number of dose groups ascended before DLT is observed, and the MTD is determined.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects voluntarily participated in the study and signed an informed consent form.
* 2.Patients with cirrhosis confirmed by histopathology, endoscopy or imaging examination without determining the etiology and in the decompensated stage.
* 3.Patients with cirrhosis that persists or progresses after adequate etiological treatment;
* 4.Model for End-Stage Liver Disease (MELD) score of 10-16 (including cut-off values).
* 5.Child-Pugh grade of liver cirrhosis is grade B (7~9 points, including the cut-off value);
* 6.Subjects with unobstructed vascular access , and who can performed peripheral blood mononuclear cell collections.
* 7.Subjects were able to communicate well with the investigator, cooperate with follow-up work, and understand and comply with the requirements of the study.

Exclusion Criteria:

* 1. Subjects who were Allergic to cell therapy, steroids, and related drugs used in the study；
* 2.At the same time, subjects who also had other uncured malignant tumors, except for local skin cancer and cervical cancer in situ that have been adequately treated and have not recurred within 5 years；
* 3.Subjects with a history of prior organ transplantation or tissue regeneration therapy；
* 4.Previously diagnosed hepatocellular carcinoma or uncertain cases (except subjects with abnormal hyperplasia or indeterminate nodules)；
* 5.Subjects with any active, known or suspected autoimmune diseases (including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enteritis, multiple sclerosis, vasculitis, glomerulonephritis, uveitis, pituitary inflammation, hyperthyroidism, etc.)；
* 6.Subjects who were systematically treated with corticosteroids (> 10 mg/day of prednisone or other equivalent hormones) or other immunosuppressants within 4 weeks prior to apheresis. In the absence of active autoimmune disease, inhaled or topical corticosteroids therapy and adrenal hormone replacement at doses ≤ 10 mg/day of prednisone efficacy are permitted；
* 7.Patients with grade 2 or above hepatic encephalopathy within 3 months prior to apheresis or current diagnosis (according to the HE grading criteria revised in the 2018 guidelines for the diagnosis and treatment of hepatic encephalopathy in liver cirrhosis);
* 8.Virology shows anti-HCV antibodies, HIV-positive, or syphilis antibodies during the screening period；
* 9.During the screening period, hepatitis B surface antigen positive (except when HBV-DNA quantification < 20 IU/mL).
* 10. Ascites or pleural effusion that cannot be controlled by appropriate intervention, those who require frequent puncture drainage (once a month or more frequently) or those who have received thoracic or ascites drainage within 2 weeks before treatment, except for a small amount of ascites or pleural effusion on imaging；
* 11.Previous or current idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis (imaging only, no hormonal therapy may be enrolled), drug-induced pneumonia, or active pneumonia on screening imaging）；
* 12.Clinical symptoms or diseases of the heart that were not well controlled, eg: (1) NYHA grade 2 or higher cardiac insufficiency, (2) unstable angina, (3) acute myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention；
* 13. Subjects with hypertension who were not well controlled by antihypertensive drugs (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥90 mmHg)；
* 14. The screening period check meets the following criteria：

  1. PLT <50 ×10*9/L；
  2. Alpha-fetoprotein was more than twice the upper limit of normal, or ALT> 5 times the upper limit of normal；
  3. Serum albumin < 30 g/L and other causes such as malnutrition or kidney disease are excluded；
  4. INR > 1.5 or PT extension more than normal +5 seconds or more。
* 15.Any of the following bleeding occurs：

  1. Previous portal hypertension bleeding；
  2. There were episodes of active bleeding that required hospitalization within 1 month prior to apheresis；
  3. History of gastrointestinal bleeding or definite gastrointestinal bleeding or bleeding events due to oesophageal and/or gastric varices within 1 month prior to apheresis；
  4. Known hereditary or acquired bleeding and thrombophilia (eg, hemophilia, coagulopathy, etc)。
* 16.Arteriovenous thrombotic events such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism occurred within 1 month before apheresis。
* 17.Anticoagulants or antiplatelet drugs were used 3 days before treatment；
* 18.Subjects had active infection within 2 weeks before apheresis, or fever of unknown origin ≥ 38.5°C within 7 days before treatment, or WBC count ≥15×109/L before apheresis, or continued antibiotics；
* 19. Pregnant and lactating women who were currently breastfeeding or are not currently breastfeeding but less than 6 months after delivery；
* 20.Female subjects (or male subjects) of childbearing age who intend to have a desire to have children during the study period (from the signing of the informed consent form) to 30 days after the end of administration and refuse to use effective contraception；
* 21.Have participated in other drug or device clinical studies within 4 weeks prior to screening；
* 22. Regular drinkers in the 1 month (30 days) prior to screening, i.e. those who drank more than 14 units of alcohol per week (1 unit = 360 beer or 45 mL of spirits or 150 mL of wine with 40% alcohol)；
* 23. According to the judgment of the investigator, the subjects had other factors that may cause the study to be terminated halfway, such as other serious concomitant diseases (such as severe diabetes, mental illness, drug use, etc.), serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subject, or the collection of data and samples；
* 24. Other factors that the investigator deemed unsuitable for inclusion or that influenced participants' participation in or completion of the study。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) Maximum Tolerated Dose (MTD) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Lianxin LX Liu, professor, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- Lianxin Liu, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No